CLINICAL TRIAL: NCT04910256
Title: The Effect of Huatuo Zaizao Pill on Neurological Function and Motor Recovery in Ischemic Stroke Patients During the Recovery Stage: a Open-labelled, Randomized Controlled Trial
Brief Title: Clinical Study on Huatuo Zaizao Pills for Post-stroke Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XiyuanH-huatuo zaizao pill
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke
Keywords: Huatuo Zaizao pill; stroke rehabilitation; limb spasticity; motor recovery; traditional Chinese medicine
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants are randomly and evenly assigned to 2 groups using block randomization.Random numbers are generated by the stratified random method using the Statistical Analysis Software （SAS） statistical software and assigned by an independent statistician at the Good Clinical Practice Institute of XiYuan Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HuaTuo ZaiZao group (Experimental): In this arm, patients take 8g of HuatuoZaizao pill three times a day. Besides，participants will receive basic treatment in accordance with the "Guidelines for diagnosis and treatment of ischemic stroke in China",and the drug and dosage will be formulated by the researchers according to the clinical situation.Treatment lasts for 12 weeks
  Interventions: Drug: Huatuo Zaizao Pills; Other: Basic treatment
- Control group (Sham Comparator): participants will receive basic treatment in accordance with the "Guidelines for diagnosis and treatment of ischemic stroke in China",and the drug and dosage will be formulated by the researchers according to the clinical situation.Treatment lasts for 12 weeks
  Interventions: Other: Basic treatment

INTERVENTIONS:
Drug: Huatuo Zaizao Pills — Patients take 8g of HuaTuo Zaizao pill three times a day. Treatment lasts for 12 weeks.
  Arms: HuaTuo ZaiZao group
Other: Basic treatment — It accordance with the "Guidelines for diagnosis and treatment of ischemic stroke in China",and the drug and dosage will be formulated by the researchers according to the clinical situation.

SUMMARY:
The purpose of this study was to evaluate the improvement of limb motor function and nerve function of patients with HTZZ during stroke rehabilitation. A total of 80 subjects will be randomly assigned to Huatuo Zaizao pill group or the control group.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled clinical trial. Eighty patients with phlegm and blood stasis block syndrome of ischemic stroke were randomly assigned to Hua Hua reconstruction group or control group at a ratio of 1:1. The treatment period is 12 weeks. The purpose is to evaluate its efficacy and safety, provide an objective basis for precise treatment of traditional Chinese medicine, and improve clinical efficacy. The main result is the changes of MAS scores 12 weeks days after taking the drug. The secondary result is the change in NIHSS, Fugl-Meyer and BI.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged between 35 and 75 years old
* 2.With a disease course between 2 weeks- 24weeks
* 3.Meeting the diagnostic criteria of ischemic stroke
* 4.Signed and dated written informed consent.
* 5.4≤NIHSS score≤22

Exclusion Criteria:

* 1.Unstable vital signs, or serious heart, liver, lung, kidney and other organ diseases
* 2.Exclude Transient Ischemic Attack(TIA)
* 3.Patients who are participating in clinical trials of other drugs within the past 1 month
* 4.Pregnant or breastfeeding women
* 5.Athletes, Epileptics, Allergic to this product

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | The change from baseline in Modified Ashworth Scale (MAS) score at week 6 and 12 [Time Frame: Baseline,6th week±3 days, 12th week±3 days]
  Modified Ashworth Scale (MAS) measure spasticity. During the administration of MAS , the examiner passively moves the joint being tested and rates the perceived level of resistance in the muscle groups opposing the movement.It is single-item measures ranging from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates that the affected part is rigid in flexion or extension.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS ) | The change from baseline in National institute of health stroke scale (NIHSS ) score at week 6 and 12 [Time Frame: Baseline,6th week±3 days, 12th week±3 days]
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item measure of the effect of acute stroke on a variety of areas including level of consciousness, neglect, motor strength, facial palsy, ataxia, dysarthria, and sensory loss.
Fugl-Meyer | The change from baseline in Fugl-Meye score at week 6 and 12 [Time Frame: Baseline,6th week±3 days, 12th week±3 days]
  The Fugl-Meyer Assessment of Sensorimotor Impairment (FM) is one of the first scales developed to quantitatively measure the recovery from hemiplegic stroke. It assesses recovery in five domains, including motor functioning of the upper and lower extremities, balance, sensation, joint range of motion, and joint pain in post-stroke patients. Each task is scored on a scale of 0-2, with 0 indicating the patient cannot perform the task and 2 indicating the patient can fully perform the task.
Barthel Index（BI） | The change from baseline in BI total score at week 6 and 12 [Time Frame: Baseline,6th week±3 days, 12th week±3 days]
  The BI is a test used in healthcare to evaluate the people's daily self care activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ding YQ, Zhao D, Chen X, Yuan HM, Mao LJ. Effect of Huatuo Zaizao Pill on Neurological Function and Limb Motor Recovery in Ischemic Stroke Patients During Convalescence: An Open-Labelled, Randomized Controlled Trial. Chin J Integr Med. 2025 Jun;31(6):483-489. doi: 10.1007/s11655-025-3928-4. Epub 2025 Apr 15. PMID 40232598